CLINICAL TRIAL: NCT04103216
Title: Development of an Effective Treatment of Cryptosporidiosis in Bangladeshi Children
Brief Title: Treatment of Cryptosporidiosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR-19079
Record Dates: First submitted 2019-09-17; First posted 2019-09-25 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Cryptosporidiosis
Keywords: Cryptosporidiosis; Treatment; Bangladesh; Nitazoxanide
MeSH Terms: conditions — Cryptosporidiosis | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: This will be a prospectively conducted randomized pilot study with 3 arms in children, where cryptosporidium infected children will receive Nitazoxanide treatment with or without the probiotic, Lactobacillus reuteriDSM 17938 and the third arm will receive the standard supportive care normally provided for Cryptosporidium infections.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention arm NItazoxanide with probiotics (Active Comparator): Child will be receive the Nitazoxanide treatment for 3 days with probiotics (L reuteri DSM 17938 ) for 7days. The doses of Nitazoxanide will be twice a day for 3 days and dosage will be 5 ml every 12 hours with food. The Nitazoxanide oral suspension contain 100mg/5ml.
  L reuteri DSM 17938 will be 2×108 CFU and will receive 5 drops orally twice daily for a consecutive 7 days.
  Interventions: Other: Nitazoxanide with Lactobacillus Reuteri DSM 17938
- Intervention arm Nitazoxanide with placebo (Placebo Comparator): Child will be receive the Nitazoxanide treatment for 3 days with placebo for 7days. The doses of Nitazoxanide will be twice a day for 3 days and dosage will be 5 ml every 12 hours with food. The Nitazoxanide oral suspension contain 100mg/5ml.
  Placebo will receive 5 drops orally twice daily for a consecutive 7 days.
  Interventions: Other: Nitazoxanide
- Control arm (No Intervention): Child will received the standard supportive care normally provided for Cryptosporidium infections

INTERVENTIONS:
Other: Nitazoxanide with Lactobacillus Reuteri DSM 17938 — Nitazoxanide with probiotics
  Arms: Intervention arm NItazoxanide with probiotics
Other: Nitazoxanide — Nitazoxanide with placebo
  Arms: Intervention arm Nitazoxanide with placebo

SUMMARY:
Background:

1. Burden:

   Cryptosporidiosis among the top 10 causes of diarrhea in the 1st year of life in low and middle-income countries (LMICs), with an estimated total of 48,000 annual deaths and accounting for 4.2 million disability-adjusted life years lost.
2. Knowledge gap:

The only approved drug for the treatment of diarrhea caused by Cryptosporidium infection is Nitazoxanide (NTZ) but NTZ has a higher failure rate in malnourished children. The lack of effective therapy for cryptosporidiosis remains an immense knowledge gap in the efforts to improve childhood health worldwide.

Hypothesis:

NTZ treatment failure in malnourished infants is due to a secondary immune deficiency that can be reversed by the appropriate therapeutic treatment. Lactobacillus reuteri DSM 17938 can have a potential immune modulating effect by altering gut microbiome promoting NTZ action.

Objectives:

Primary:

• To develop new approaches to treat and prevent cryptosporidiosis

Secondary:

* Determination of the treatment outcome of NTZ against cryptosporidiosis in Bangladeshi children.
* Determination of the change in effectiveness of NTZ treatment in conjunction with the administration of probiotics in malnourished Bangladeshi children with cryptosporidiosis

Methods:

This will be a prospectively conducted randomized pilot study with 2 arms in children in the Mirpur (Dhaka, Bangladesh) slum area, where cryptosporidium infected children will receive Nitazoxanide treatment with or without the probiotic, Lactobacillus reuteri DSM 17938.

Outcome measures/variables:

The significance of the work lies in the ability of the study to provide new approaches to treat and prevent Cryptosporidiosis. The goal of this work is to assess the efficacy of NTZ drug in a low socioeconomic Bangladeshi population and establish new supportive therapeutic measures to the already established treatment with NTZ against in cryptosporidiosis.

DETAILED DESCRIPTION:
Background: Reports from longitudinal birth cohort study at Bangladesh show that 77% of children experience at least one incidence of cryptosporidiosis in the first two years of life. Cryptosporidiosis is also associated with the development of malnutrition leading to an estimate of an additional 4.2 million disability adjusted life years lost. A number of studies on cryptosporidiosis conducted at icddr,b showed that Cryptosporidium sp. was one of the most important causative agents of diarrhea associated with morbidity and mortality. Previous studies at icddr,b also made a number of other intriguing elucidations, which include:

1. Cryptosporidium sp. infected most children in the 1st year of life in a cohort at Mirpur, Dhaka. Investigators observed that up to 64% of infants were diagnosed with cryptosporidiosis in the 1st year of life while 26% of these cases had accompanying co-infections.
2. Cryptosporidium sp. was established as a top 10 diarrheal pathogen, with infections occurring with multiple other enteropathogens. Investigators discovered that infection and diarrhea with multiple entero-pathogens in infants in an LMIC setting was the norm, without any exception. On average each infant in Mirpur, Bangladesh had 3-5 enteric pathogens present in their stool at any a single time point.The importance of Cryptosporidium as a leading cause of infant diarrhea was validated by the MAL-ED study conducted across 8 different low to middle income sites.
3. Diarrhea due to Cryptosporidium in the first year of life was independently associated with the future development of malnutrition.
4. Impaired neurocognitive development at two years of age for infants with history of cryptosporidiosis as measure using the Bayley's scales of infant development.

Currently, there is no effective vaccine for cryptosporidiosis and the only approved drug for the treatment of diarrhea caused by Cryptosporidium infection is nitazoxanide (NTZ)(U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES 2003). NTZ is the only treatment but its efficacy in controlled clinical trials has varied widely. While this drug has been generally shown to have an efficacy of >80%, in previous studies involving malnourished Zambian children it was shown to have an efficacy of only 56%. An effective therapy would be appealing for cryptosporidiosis in children in the developing world where the burden of infection is high and where persistence of the enteropathogen in the absence of diarrhea is associated with malnutrition.

Although the exact reason for NTZ exhibiting a higher failure rate in malnourished children is unclear, this drug has been shown to inhibit the pyruvate-ferredoxin oxidoreductase of parasites and anaerobic bacteria but its effectiveness in combating cryptosporidiosis is dependent on the host immune competence. The gut micro-environment is a key component of the host response to environmental challenge, with the gut microbiota being postulated to mediate integral roles in promoting and calibrating all aspects of the immune system. Fermented products (such as yogurt) have long been thought to promote health. However, in most commercial food products the levels of the beneficial microorganisms or probiotics are not consistent and at lower levels than required for the desired biological effect. Lactobacillus reuteri DSM 17938 has been one of the most extensively studied probiotic in children and adults with functional gastrointestinal disorders. Lactobacillus reuteri DSM 17938 in particular would be effective against cryptosporidiosis due to the presence of both microorganisms at duodenum of human. A recent study at icddr, b has shown this commonly used probiotic appeared safe and well-accepted by Bangladeshi families. Lactobacillus reuteri has been tested in clinical trials and has attained the "GRAS (generally regarded as safe)" status for use in both children and adults and has additionally demonstrated immunomodulatory activities. This probiotic is thus hypothesized to act as a beneficial supplement to the NTZ treatment in cryptosporidiosis through a potential reduction in the gut inflammation resulting from Cryptosporidium infection. Additionally, if the microbiota treatment promotes parasite clearance and decrease the burden, it will be associated with faster disease resolution and better clinical outcomes. Lactobacillus reuteri DSM 17938 has been reported to inhibit the RORa/y activity to suppress Th17 cells, thus promoting an appropriate immune response in improving the efficacy of the drug treatment. The Probiotic VSL#3 which contains Lactobacillus reuteri DSM 17938 as well as other bacteria with anti-inflammatory activities has been shown to reduce the severity of inflammatory diarrhea in animal models and has been included as one of the treatment options for pouchitis by the British Society of Gastroenterology. Investigator's goal in this study is to undertake an iterative approach to improve and optimize the currently used most effective treatment regime against cryptosporidiosis.

Experimental Design and Methodology:

The objectives of the study are to investigate 1) Determine the incidence of Cryptosporidiosis 2) Assessment of the acquired immune response to Cryptosporidiosis and 3) Analyze the human genes influencing susceptibility to Cryptosporidiosis. The proposed study will utilize the field setting of the parent study. This proposed pilot study will help to elucidate the effective treatment for cryptosporidiosis which will not only help the study participants of the parent study, but also help other individuals with cryptosporidiosis from similar settings. Later on the parent study findings will provide information which will help to investigate host immune mechanism and permit the design of new strategies incorporating host-directed therapies that could optimize an appropriate immune response improving the efficacy of the NTZ with probiotics treatment.

Study products: Nitazoxanide will be purchased from local commercial Square pharmaceuticals Ltd. and probiotics will be purchased from Bio Gaia a Swedish health care company.

Study details: This will be a randomized clinical trial to be conducted prospectively in a pilot scale. The study will be conducted at Mirpur (Dhaka, Bangladesh) slum areas. The parent organization maintains a field site for studies on cryptosporidiosis. This is an area with a high incidence of both cryptosporidiosis and child malnutrition. Identified participants will be screened by strict maintenance and following of the inclusion and exclusion criteria. The study staff will take consent from the patient's legal guardian to enroll the child. Investigators will screen 975 children presenting age 12 months to 36 months, of either sex and having no history of antibiotic use in the last month before enrollment. The prevalence of Cryptosporidium infection in the proposed age group in that community is approximately 8%. Investigators will enroll 78 participants with cases of Cryptosporidiosis, diagnosed using animmune assay from stool. Investigators will enroll both symptomatic and asymptomatic children. Study physician will collect all the demographic, socioeconomic, anthropometric, clinical and treatment information. A random number generator will be used to determine which treatment group to which the child will be assigned. Stool and anthropometric information will be collected from all groups onenrollment, on day 4 (day after NTZ treatment), on day 8 (day after Probiotics treatment), on day 90 (follow-up on 3 months) and on day 180 (follow-up on 6 months). Rate of decrease of oocyst load by qPCR in stools at Days 4 and day 8 will be tested.

Study Schedule: Complete study schedule details listed by study visit are described below.

Enrollment

* Taking of informed consent
* Anthropometric measurement
* Enrollment questionnaire
* Stool collection for immune assay of the detection of cryptosporidiosis and quantitative PCR for the baseline parasites load

Start of Intervention (Day 1)

* Review of eligibility of enrollment
* Anthropometric measurement
* Start the intervention

Visit Day 2 and 3

* Administration of intervention
* Screening for adverse events

Visit Day 4

* Administration of intervention
* Screening for adverse events
* Stool collection for q PCR

Visit Day 5, 6 and 7

* Administration of intervention
* Screening for adverse events

Visit Day 8

* Screening for adverse events
* Stool collection for q PCR

Visit Day 20

* Screening for adverse events
* Stool collection for q PCR

Follow up visit day 90 and 180

* Anthropometric measurement
* Stool collection

Intervention:Child will be randomly selected to receive either the NTZ treatment for 3 days with probiotics for 7days or the NTZ treatment for 3 days with placebo for 7days or to receive the standard supportive care normally provided for Cryptosporidium infections. The doses of NTZ will be twice a day for 3 days and L reuteri DSM 17938 will be 2×10^8 CFU will be taken orally. Treatment group will receive 5 drops probiotic twice daily for a consecutive 7 days and placebo group will receive NTZ for 3 days without probiotic. The NTZ dosage will be 5 ml every 12 hours with food. The NTZ oral suspension contain 100mg/5ml.

This drug NTZ and probiotics usually has no side effects. Prior study suggests no adverse event or serious adverse event.

Expected drop-out: From previous experience the drop-out rate is very low. Investigator considered 10% drop out in each group.

Sample size: This will be a pilot study with a total of 105 patients distributed equally across the three above mentioned study arms. A sample size of N = 105 individuals (35 in each of the groups) will be sufficient to detect a clinically important difference of the proportion (at least) 24% between the groups, using a two-sided Z-test of the difference between proportions with 80 % power and a 5 % level of significance and a precision of 0.10. This 24 % difference represents the difference between the prevalence of 56% in the NTZ+placebo group and 80 % in the NTZ+probiotics group. With consideration of 10% attrition rate, the total sample size is 117 individual (39 in each group). Since this is a pilot study and due to small funding, the precision value considered 0.10.

Data analysis plan: Database will be created after getting the lab test values. Data will be analyzed using SPSS (version 16). Treatment efficacy will be measured in three groups. Nature of data distribution will be checked whether it is normally distributed or not. Using two sample mean test among group will be compared using parametric (t-test) or non-parametric (Mann-Whitney test) where applicable. Investigator will be examined, if there is any difference in cryptosporidium infection outcome of treatment with NTZ+placebo in comparison NTZ+probiotics treatment in children and then paired parametric-test or paired non-parametric test will be done depending on data distribution. Investigator will also examine the treatment effectiveness in malnourished children. Multivariate logistic regression will be performed to examine the effect of socioeconomic condition, nutrition and other clinical conditions associated with different treatment on cryptosporidiosis.

ELIGIBILITY:
Inclusion Criteria:

• Children will be enrolled with cryptosporidium infection positive from Mirpur, Dhaka, Bangladesh and whose parents or legal guardian will give consent.

Exclusion Criteria:

* Participants with history of prior antibiotic use before enrollment
* Participants suffering from Severe Acute Malnutrition, with a WHO median weight for length Z score (WLZ) of less than -3 or having bilateral pedal edema).

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
To develop new approaches to treat and prevent cryptosporidiosis | Change from baseline cryptosporidium oocyst load at day 8.
  Cryptosporidium infection outcome of treatment with Nitazoxanide and probiotics in comparison Nitazoxanide treatment in children. Change from baseline cryptosporidium oocyst load in stools at day 8 will be tested by qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Zannatun Noor, PhD, Principal Investigator — Assistant Scientist, Infectious Diseases Division, icddr,b
Locations (1):
- Icddr,B, Dhaka, Bangladesh